CLINICAL TRIAL: NCT04939558
Title: A Longitudinal Observational Study to Investigate the Patterns of Change in the Tidal Breathing CO2 Waveform, Measured Using the N-Tidal C Handset, in Patients With COPD Compared to Patients With Other Common Cardiorespiratory Conditions
Brief Title: Cardiorespiratory Diagnostic Study
Acronym: CARES
Status: Completed | Type: Observational
Sponsor: TidalSense (Industry)
Collaborators: Innovate UK (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: G001-21
Record Dates: First submitted 2021-06-03; First posted 2021-06-25 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: COPD; Asthma; Lung Cancer; Anemia; Congestive Cardiac Failure; Bronchiectasis; Interstitial Lung Disease; Long COVID; Upper Respiratory Disease; Healthy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Lung Neoplasms; Anemia; Heart Failure; Bronchiectasis; Lung Diseases, Interstitial; Post-Acute COVID-19 Syndrome; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Chronic Obstructive Pulmonary Disease: 245 participants - GOLD 1, 2, 3 / A, B, C
  Interventions: Device: N-Tidal C handset
- Asthma: 55 participants - Mild to moderate, not labelled as severe.
  Interventions: Device: N-Tidal C handset
- Congestive cardiac failure: 55 participants
  Interventions: Device: N-Tidal C handset
- Anaemia: 55 participants - with at least 50% of participants recruited having no history of chronic cardiorespiratory conditions
  Interventions: Device: N-Tidal C handset
- Bronchiectasis: 55 participants - Acquired or genetic, e.g. cystic fibrosis or other primary ciliary dyskinesias
  Interventions: Device: N-Tidal C handset
- Lung cancer: 55 participants - including rare types e.g. mesothelioma
  Interventions: Device: N-Tidal C handset
- Interstitial Lung Disease: 55 participants - including pulmonary fibrosis pneumoconiosis, asbestosis, sarcoidosis, amyloidosis
  Interventions: Device: N-Tidal C handset
- Long COVID: 55 participants
  Interventions: Device: N-Tidal C handset
- Upper airway obstruction disorder: 55 participants
  Interventions: Device: N-Tidal C handset
- Healthy: 55 participants - with no previous or current chronic cardiorespiratory diagnoses
  Interventions: Device: N-Tidal C handset

INTERVENTIONS:
Device: N-Tidal C handset — Participants are to use the 'N-Tidal C' handset every day for 14 days. This will ideally be two times a day (once in the morning and once in the evening, before using any regular inhalers). Each breath record requires the participant to breathe through the mouthpiece for 75 seconds in a relaxed manner.

SUMMARY:
This study uses a new breathing device called 'N-Tidal C' handset which measures breathing patterns. Investigators have found that people with cardiac and respiratory illnesses breathe out a gas, called carbon dioxide (CO2), in a different way to healthy people. The pattern of breathed out CO2 (the waveform) varies according to the underlying health of the user's lungs. Monitoring these changes may help doctors to more accurately diagnose and monitor the most common and serious respiratory conditions.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is among the most prevalent respiratory conditions, and in the top five causes of death worldwide. However, mis-diagnosis rates are high (both under- and over- diagnosis), owing to the lack of a simple, reliable and specific diagnostic test. In addition, COPD is often diagnosed late in the natural history of the disease, which misses the opportunity for early intervention, with early treatment and health-behaviour changes (smoking cessation).

Spirometry, the current gold standard for diagnosis, is unreliable (technique-dependent), crude (measures airflow), and non-specific (multiple respiratory conditions can produce similar patterns on spirometry). It also relies on proper administration by specially trained members of staff. As a result, spirometry is often (a) not performed before a speculative diagnosis of COPD is made, and (b) performed poorly, resulting in poor-quality information on which to base a respiratory diagnosis.

There is therefore a need for a simple, reliable, robust and accurate test for diagnosing COPD which is non-operator dependent, and non-technique dependent.

Currently, capnography is invasive, expensive and can only be recorded in specialist centres via a nasal cannula and micro-stream sampling of expired carbon dioxide in the intensive care setting. The N-Tidal C (NTC) handset, a new (CE-marked), hand-held, wireless device has been developed to monitor the user's Tidal Breathing CO2 (TBCO2) waveforms at rest, during normal tidal breathing. This device can be safely operated in the home environment, has a battery life of weeks, and has an isolated, disposable, breath pathway that isolates an individual's breath from the rest of the device, making it safe to reuse between patients after the outer casing has been decontaminated using a 3-stage disinfection process.

The N-Tidal technology has the potential to offer new insights into lung physiology (above and beyond those currently available from spirometry and lung function testing), and early evidence from TidalSense's previous clinical studies suggests that the TBCO2 data could be used to fingerprint and diagnose COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Healthy volunteer (with no previous or current chronic cardiorespiratory diagnoses)

One of the following cardiorespiratory diagnoses:

* COPD (GOLD 1, 2, 3 / A, B, C)*
* Asthma (mild to moderate, not labelled as severe)*
* Congestive cardiac failure*
* Anaemia (with at least 50% of participants recruited having no history of chronic cardiorespiratory conditions)*
* Bronchiectasis (acquired or genetic, e.g. cystic fibrosis or other primary ciliary dyskinesias)*
* Lung cancer (including rare types e.g. mesothelioma)*
* Interstitial Lung Disease (including pulmonary fibrosis pneumoconiosis, asbestosis, sarcoidosis, amyloidosis)*
* Long COVID*
* Upper airway obstruction disorder*
* [Active pulmonary hypertension]
* [Extrinsic Allergic Alveolitis]
* [Active pulmonary embolism]

Exclusion Criteria:

* Participants who, in the opinion of the chief investigator, or their delegate, are unlikely to comply with the requirements of the study;
* Diagnosis of neuromuscular disorders;
* Concurrent diagnosis of cardiorespiratory conditions (other than those listed in the inclusion criteria above) that, in the opinion of the chief investigator, would impact the conduct of the study
* Participants who are acutely unwell, e.g. active exacerbation, very short of breath e.g. severe COPD (GOLD 4 / D) or end-stage IPF.
* Inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from among the primary care patient population served by the Modality (GP) partnership. Participants will either be healthy (no underlying cardiorespiratory diagnoses) or have one of the following conditions: COPD, asthma, congestive cardiac failure (heart failure), bronchiectasis (including cystic fibrosis), anaemia, lung cancer (including mesothelioma), pulmonary fibrosis, long COVID, an upper airway obstruction disorder, pulmonary embolism, pulmonary hypertension, extrinsic allergic alveolitis.
  Participants will deliberately be recruited from a wide range of demographic backgrounds, to provide diversity of: age, gender, geographic location and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Breath records from participants with Chronic Obstructive Pulmonary Disease (COPD) | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 245 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 6860 records

SECONDARY OUTCOMES:
Breath records from Healthy volunteers (no previous or current cardiorespiratory diagnoses) | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Asthma | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Congestive cardiac failure | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Anaemia | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Bronchiectasis | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Lung cancer | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Interstitial Lung Disease | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Long COVID | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records
Breath records from participants with Upper airway obstruction disorder | 12 months from First Patient First Visit (FPFV)
  Tidal Breathing CO2 waveform data from 55 participants collected using the N-Tidal C Handset.
  Each participant delivering 2 x breath records per day for 14 days = 1540 records

CONTACTS AND LOCATIONS:
Overall Officials: Zishan Ali, MBBS BSc, Principal Investigator — Modality Partnership; Elango Vijaykumar, MBBS, FRCG, Principal Investigator — Modality Partnership
Locations (1):
- Modality Partnership, Birmingham, West Midlands, United Kingdom